CLINICAL TRIAL: NCT06422767
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Bepirovirsen on Cardiac Conduction as Assessed by 12-lead Electrocardiogram in Healthy Volunteers
Brief Title: Study to Evaluate the Effect of Bepirovirsen on Cardiac Conduction as Assessed by 12-lead Electrocardiogram in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205873
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis B
Keywords: Bepirovirsen; Cardiac Conduction; Electrocardiogram; QT interval corrected by Fridericia's formula; Hepatitis B virus
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Bepirovirsen (Experimental)
  Interventions: Drug: Bepirovirsen
- Participants receiving Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bepirovirsen — Bepirovirsen will be administered.
  Arms: Participants receiving Bepirovirsen
Drug: Placebo — Placebo will be administered.
  Arms: Participants receiving Placebo

SUMMARY:
This study will evaluate the effect of a single dose of bepirovirsen on the QT interval corrected by Fridericia's formula (QTcF) as compared to placebo. The data generated will be used to model the relationship between bepirovirsen concentration and QTcF.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, electrocardiogram (ECG) and vital signs.
* Body weight greater than equal to (>=) 50 Kilograms (kg) and Body mass index (BMI) within the range 19-32 Kilograms per square meter (kg/m^2) (inclusive).
* Study will enroll both male and female participants.

  o Female participants are eligible to participate if they are not pregnant or breastfeeding and are either not of childbearing potential or agree to using a highly effective method of contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* History of vasculitis or presence of symptoms and signs of potential vasculitis
* History of lymphoma, leukemia, or any malignancy except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for at least 3 years.
* Participants with any other medical conditions which, in the judgement of the investigator and/or Medical Monitor, could jeopardize the integrity of the data derived from that participant or the safety of the participant.
* Past, current or intended use of over-the-counter or prescription medication, including herbal medications within 7 days or 5 half-lives (whichever is longer) before dosing.
* Current or recent use of creatine-containing supplements, or intended use up to 50 days post-dosing.
* Prior treatment with any oligonucleotide or small interfering Ribonucleic acid (RNA) (siRNA) within 12 months before dosing.
* Exposure to more than 4 new chemical entities within 12 months before the first dosing day
* Current enrollment or past participation in another investigational study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered within 5 half-lives (if known) or twice the duration of biological effect (if known), whichever is longer, or within the last 90 days (if half-life and duration of biological effect are unknown), before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Current enrollment or past participation in this clinical study.
* Positive pre-clinical drug/alcohol screen, including tetrahydrocannabinol.
* Positive Human Immunodeficiency Virus antibody test.
* History or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* Regular alcohol consumption within 6 months prior to screening defined as an average weekly intake of >14 units for males or females.
* Regular use of known drugs of abuse, including tetrahydrocannabinol.
* Sensitivity to heparin or history of heparin-induced thrombocytopenia.
* History of sensitivity to bepirovirsen or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor contraindicates their participation.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Positive test results for Hepatitis B surface antigen (HBsAg), hepatitis C antibody or hepatitis C RNA at screening or within 3 months prior to first dose of study intervention.
* Known history of heart disease, including ischemic heart disease, cardiomyopathy, clinically significant cardiac arrhythmias, clinically significant valvular disease, or hypertensive heart disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in QT interval corrected by Fridericia's formula (QTcF) | Baseline (Day 1) and up to Day 4

SECONDARY OUTCOMES:
Change from Baseline in heart rate (HR) using by-time point analysis | Baseline (Day 1) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 27, 30, 33, 36, 48, 51, 54, 57, 60 and 72 hours post-dose
Change from Baseline in QT interval, corrected by Fridericia's formula (QTcF), using by-time point analysis | Baseline (Day 1) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 27, 30, 33, 36, 48, 51, 54, 57, 60 and 72 hours post-dose
Change from Baseline in PR interval using by-time point analysis | Baseline (Day 1) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 27, 30, 33, 36, 48, 51, 54, 57, 60 and 72 hours post-dose
Change from Baseline in QRS duration using by-time point analysis | Baseline (Day 1) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 27, 30, 33, 36, 48, 51, 54, 57, 60 and 72 hours post-dose
Number of participants with outlier results for QT interval, corrected by Fridericia's formula (QTcF), HR, PR and QRS | Up to Day 4
Number of participants with treatment emergent changes of T wave morphology and U-wave presence | Up to Day 4
Plasma concentrations of Bepirovirsen | Up to Day 4
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) of Bepirovirsen | Up to Day 4
Area under the concentration-time curve from time zero (pre-dose) to 24 hours post-dose (AUC[0-24]) of Bepirovirsen | Up to 24 hours
Maximum concentration (Cmax) of Bepirovirsen in plasma | Up to Day 4
Time to reach Cmax (Tmax) of Bepirovirsen | Up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/